CLINICAL TRIAL: NCT06947083
Title: Phase II Study of Elranatamab as Maintenance Therapy Post Ciltacabtagene-autoleucel(Cilta-cel) in Patients With Clinical High Risk Relapsed Myeloma
Brief Title: Elranatamab Post Cilta-cel in Patients With Clinical High Risk Relapsed Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23564
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elranatamab Maintenance Therapy (Experimental): Patients who have received cilta-cel without evidence of disease progression and have clinical high-risk myeloma, will be treated with Elranatamab as maintenance therapy for a total of 12 months starting 3-6 months post cilta-cel infusion, at the FDA approved full dose.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Maintenance therapy

SUMMARY:
The purpose of the study is to evaluate the effect of Elranatamab therapy after cilta-cel measuring how long a patient with high risk relapsed myeloma lives without the myeloma getting worse(progressing), also known as progression-free survival (PFS). Patients with clinical high-risk myeloma, defined as having history of myeloma that has grown outside of the bones or having high risk mutations in the myeloma cells, benefit less from cilta-cel compared to myeloma patients without these characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Have received commercial cilta-cel within 3-6 months for relapsed refractory myeloma and have high risk cytogenetics by IMW (del17p, or t(4;14) or t(14;16) or history of EMD, and must not have evidence of progressive disease by IMWG criteria(Appendix B) following CAR-T cell therapy.
* Have received >2 prior treatment regimens including an immunomodulatory drug, a proteasome inhibitor and a CD38 monoclonal antibody.
* Able to adhere to the study visit schedule and other protocol requirements.
* Patients must have available clonoseq ID prior to enrollment to track MRD status.
* Eastern Cooperative Group (ECOG) Performance Status of 0 or 1.
* Serum bilirubin levels ≤1.5 times the upper limit of the normal range for the laboratory (ULN), unless related to Gilbert syndrome.
* Serum AST or serum ALT levels ≤2 x ULN.
* Must have adequate bone marrow function.

Exclusion Criteria:

* Ongoing active infection defined as an infection that is worsening despite therapy and causing symptoms or requiring intravenous antibiotic treatment.
* Ongoing CRS or ICANS of any grade.
* Active plasma cell leukemia.
* Patients with CNS involvement, including meningeal involvement.
* Patients with history of Guillain-Barre syndrome.
* Uncontrolled medical problems such as diabetes mellitus, congestive heart failure, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma, which in the opinion of the treating physician pose an unacceptable risk to the patient.
* Pregnant or lactating females.
* Concurrent use of other anti-cancer agents or treatments.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible. Note: patients with hepatitis C previously treated with curative intent are considered eligible.
* Patients with renal failure requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Surival (PFS) | Up to 24 Months
  Progression-free survival (PFS) is measured from the date of initiation of Elranatamab (i.e., on-treatment date) to either the date of death from any cause or the date of disease progression, whichever comes first.

SECONDARY OUTCOMES:
Complete Response | Up to 12 months
  Proportion of participants with a complete response at the end of treatment.
MRD Negative | Up to 12 months
  Proportion of participants with MRD negativity at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided